CLINICAL TRIAL: NCT07243340
Title: A Phase I/IIa Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of Herpes Virus C5252 Injection in Patients With Intracranial Tumor
Brief Title: A Phase I/IIa Study of C5252 in Patients With Intracranial Tumor
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-C5252-003
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Glioma, Malignant
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Herpes Virus C5252 Injection (Experimental)
  Interventions: Biological: Herpes Virus C5252 Injection

INTERVENTIONS:
Biological: Herpes Virus C5252 Injection — C5252 will be administered at designed dose level.

SUMMARY:
This study includes phase I dose escalation part and phase IIa dose expansion part. The goal of this clinical trial is to learn if C5252 treatment is safe and well tolerated in patients with intracranial tumor and to learn preliminary efficacy of C5252. In this study, participants will be given single or multiple doses of C5252 according to protocol followed by toxicity observation, safety follow-up and long-term follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed recurrent malignant high-grade (WHO grade 3-4) glioma who have received standard therapy and no available treatment.
* Measurable lesions exist in accordance with RANO criteria.
* Sufficient space for ≥1 mL drug infused into tumor cavity post resection.
* Ommaya reservoir has been placed in the operation area, and drug administration conditions are available.
* Karnofsky Performance Status (KPS) ≥ 60%
* Life expectancy > 12 weeks.
* No severe hematological, cardiovascular, liver or kidney diseases.
* If the patient is a sexually active female of childbearing potential or if the patient is a sexually active male whose partner is a female of childbearing potential, the patient must use appropriate contraceptive measures for the duration of the treatment and for 6 months afterwards. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days of before the C5252 infusion.
* Capable of understanding and complying with protocol requirements.

Key Exclusion Criteria:

* Inability to undergo MRI examination for any reason.
* Active hemorrhage observed before enrollment.
* Imaging test: a. lesion located in non-cerebral regions; b. there are other lesions outside target tumor cavity; c. extra-cranial metastasis.
* Tumor lesion locates in ventricular system or there is a clear perforation between the tumor cavity and the ventricle after tumor resection.
* History of encephalitis, multiple sclerosis or other central nervous system infections
* Treated with steroid hormones and/or more than 5 mg dexamethasone per day or other immunosuppressive drugs for systemic treatment within 4 weeks.
* Persistent or active infection, and cannot be controlled by treatment.
* Subjects with bleeding tendency or need to take anticoagulant drugs, antiplatelet drugs or non-steroidal anti-inflammatory drugs (NSAIDs) and are unable to discontinue.
* Uncontrolled disease, including but not limited to symptomatic congestive heart failure, unstable angina pectoris.
* Other malignant tumor within 5 years.
* Patients who require an attenuated or live vaccine within 28 days prior to the first trial drug administration and during the study treatment period.
* In the period of recurrent herpes simplex virus infection, with corresponding clinical manifestations.
* Systemic use (other than topical) of anti-HSV drugs
* Prior treatment with any oncolytic virus, cell therapy or gene therapy.
* Participants have a history of splenectomy, organ transplantation, bone marrow transplantation or stem cell transplantation
* Prior antitumor treatment with intracranial implants, such as Carmustine.
* Previous history of allergic reactions to similar biological components such as HSV-1, IL-12 or anti-PD-1 antibodies, or with known allergic reactions to any component of the C5252 prescription, including glycerol.
* Developed ≥Grade 3 irAE during previous immunotherapy
* History of frequent drug use (including "recreational use") or drug abuse (including alcohol abuse) within one year prior to signing the informed consent form.
* Other situation that PI consider subjects not appropriate to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of adverse event | Up to 30 days after completion of treatment
  TEAE, SAE, DLT, AESI during treatment period
Phase I: Determine the MTD/RP2D | up to 4 weeks
  Maximal Tolerated Dose/Recommended Phase 2 Dose (MTD/RP2D)
Phase II: Overall Survival | Up to 2 years
  The overall survival for each patient receiving C5252 will be calculated.
Phase II: OS rate | Up to 2 years after first dose
  OS rate at 6, 12, 18 and 24 months after first study dose

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality, China